CLINICAL TRIAL: NCT05136924
Title: A Randomized, Controlled, Double-Masked, Two-Arm Investigator-Initiated Study to Assess the Efficacy of OC-01 (Varenicline) Nasal Spray on Signs and Symptoms of Dry Eye Disease in Subjects Following Corneal Collagen Crosslinking (CXL)
Brief Title: IIT Assessing OC-01Nasal Spray on Symptoms of DED Following CXL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Vance Thompson Vision - MT (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: The CIrCles Study
Record Dates: First submitted 2021-10-07; First posted 2021-11-30 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Varenicline; Nasal Sprays

STUDY DESIGN:
Intervention Model Description: OC-01 (varenicline 1.2mg/ml) nasal spray Or Placebo (vehicle) nasal spray
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A Randomized, Controlled, Double-Masked, Two-Arm Investigator-Initiated studyOC-01 (varenicline 1.2mg/ml) nasal spray Or Placebo (vehicle) nasal spray
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- OC-01 (Experimental): (varenicline 1.2mg/ml) nasal spray
  Interventions: Drug: OC-01 (varenicline 1.2mg/ml) nasal spray vs Placebo
- Placebo (Placebo Comparator): (vehicle) nasal spray
  Interventions: Other: Placebo (vehicle) nasal spray

INTERVENTIONS:
Drug: OC-01 (varenicline 1.2mg/ml) nasal spray vs Placebo — OC-01 nasal spray containing varenicline for treatment of signs and symptoms of DED. OC-01 (varenicline) nasal spray activates the trigeminal parasympathetic pathway and stimulates natural tear production to bathe the corneal nerve endings in a protective layer of tear film. In addition, OC-01 (varenicline) acts as a cholinergic agonist and may provide analgesia by activating the trigeminal parasympathetic pathway VS Placebo
  Other Names: Placebo (vehicle) nasal spray
  Arms: OC-01
Other: Placebo (vehicle) nasal spray — Placebo (vehicle) nasal spray
  Arms: Placebo

SUMMARY:
A Randomized, Controlled, Double-Masked, Two-Arm Investigator-Initiated study to Assess the Efficacy of OC-01 (varenicline) Nasal Spray on signs and symptoms of Dry Eye Disease in subjects following Corneal Collagen Crosslinking (CXL)

DETAILED DESCRIPTION:
Rationale for Study Design This study is a single center, prospective, randomized, controlled, double-masked, two-arm investigator-initiated study to investigate the efficacy of OC-01 on signs and symptoms of dry eye disease in subjects following corneal collagen crosslinking (CXL).

2. STUDY OBJECTIVES 2.1 Primary Objective

* Mean change in NEI VFQ-25 from baseline to Day 0, Day 7, and Day 28 (1-month postoperative CXL)
* Coneal epithelial healing rate at days 2 (48 hours), 3 (72 hours), 4 (96 hours) after creation of 9 mm corneal epithelial defect as evaluated by masked physician 2.2 Secondary Objectives
* Mean change in eye dryness score (EDS) as measured by the Visual Analogue Scale (VAS) from baseline overtime to Day 28 (1 month postoperatively CXL) as measured by masked evaluator
* Mean change in corneal fluorescein staining from baseline to Day 0 (surgical day) and Day 0 to Day 28 (1-month postoperative CXL) as evaluated by masked physician
* Mean change in tear break up time (TBUT) from baseline to Day 0 (surgical day) and day 0 to day 28 (1-month postoperative CXL)
* Incidence and severity of adverse events

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to sign the informed consent form

  * Be at least 18 to 50 years of age at the screening visit
  * Have best corrected manifest refraction between 20/40 to 20/100
  * Remove contact lenses 2 weeks prior to surgical procedure and continue until end of study with the exception of scleral lens wearers that have no better option for correcting visual acuity
  * Have planned corneal collagen crosslinking for treatment of keratoconus or corneal ectasia
  * Be literate and able to complete questionnaires independently
  * Be able and willing to use the study drug and participate in all study assessments and visits Have sufficient hand strength, in the opinion of the Investigator, to be able to independently administer the study drug
  * Have provided verbal and written informed consent
  * If a female is of childbearing potential, they must: use an acceptable means of birth control (acceptable methods of contraception include: hormonal - oral, implantable, injectable, or transdermal contraceptives, mechanical - spermicide in conjunction with a barrier such as a diaphragm or condom, IUD, or surgical sterilization of partner), and have a negative urine pregnancy test on Baseline/Screening Day

Exclusion Criteria:

* Have presence of corneal pathology that may interfere with CXL outcomes

  * At time of screening have had temporary plugs placed in the past 1 month or currently have permanent punctal plugs in place
  * Active infectious, ocular, or systemic disease
  * Have a history of ocular inflammation or macular edema
  * Have chronic or recurrent epistaxis, coagulation disorders or other conditions that, in the opinion of the Investigator, may lead to clinically significant risk of increased bleeding
  * Have had nasal or sinus surgery (including history of application of nasal cautery) or significant trauma to these areas
  * Have a vascularized polyp, severely deviated septum, chronic recurrent nosebleeds, or severe nasal obstruction as confirmed by intranasal examination performed at Visit 1.
  * Be currently treated with nasal continuous positive airway pressure
  * Have had blepharoplasty in either eye
  * Have had a corneal transplant in either eye
  * Have a history of seizures or other factors that lower the subject's seizure threshold.
  * Have a systemic condition or disease not stabilized or judged by the Investigator to be incompatible with participation in the study or with the lengthier assessments required by the study (e.g., current systemic infection, uncontrolled autoimmune disease, uncontrolled immunodeficiency disease, history of myocardial infarction or heart disease, etc.)
  * Have a known hypersensitivity to any of the procedural agents or study drug components Have current concomitant use of a nicotinic acetylcholine receptor agonist [Nicoderm®, Nicorette®, Nicotrol NS® (nicotine), Tabex®, Desmoxan® (cytisine), and Chantix® (varenicline)] within the previous 30 days of Visit 1 and during the treatment period.
  * Have active or uncontrolled, severe (at the discretion of the investigator):

    * Systemic allergy
    * Chronic seasonal allergies at risk of being active during the study treatment period
    * Rhinitis or sinusitis requiring treatment such as antihistamines, decongestants, oral or aerosol steroids at the Screening Visit or be expected to require treatment during the treatment period of the study
  * Untreated nasal infection at Visit 1
  * Have any condition or history that, in the opinion of the investigator, may interfere with study compliance, outcome measures, safety parameters, and/or the general medical condition of the subject
  * Be currently enrolled in an investigational drug or device study or have used an investigational drug or device within 30 days prior to Visit 1 and during the treatment period.
  * Be a female who is pregnant, nursing, or planning a pregnancy at Visit 1. Be a woman of childbearing potential who is not using an acceptable means of birth control; acceptable methods of contraception include: hormonal - oral, implantable, injectable, or transdermal contraceptives; mechanical - spermicide in conjunction with a barrier such as a diaphragm or condom; IUD; or surgical sterilization of partner.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
NEI VFQ-25 Questionnaire | from baseline to Day 28 (1-month postoperative CXL)
  questionnaire assesses effect of visual impairment on the patient's current health-related quality of life, including questions dealing with irritation in and around the eye. The score on a scale is from 0 to 100 points. A score of 0 is the worst score and a score of 100 is the best score and means the patient has no vision problems
Corneal Epithelial Healing | Up to 96 hours after creation of 9mm epithelial defect
  Corneal epithelial healing rate at days 2 (48 hours), 3 (72 hours), 4 (96 hours) after creation of 9mm epithelial defect as measured by a masked physician

SECONDARY OUTCOMES:
Dryness Scoring | from baseline over time to Day 28 (1 month postoperatively CXL)
  Mean change in eye dryness score (EDS) as measured by the Visual Analogue Scale (VAS) from baseline over time to Day 28 (1 month postoperatively CXL) as measured by masked evaluator
Corneal Fluorescein Staining | from baseline to Day 0 (surgical day) and Day 7 to Day 28 (1-month postoperative CXL)
  Mean change in corneal fluorescein staining from baseline to Day 0 (surgical day) and Day 7 to Day 28 (1-month postoperative CXL) as evaluated by masked physician
Tear Break Up Time | baseline to Day 0 (surgical day) and Day 7 to Day 28 (1-month postoperative CXL)
  Mean change in tear break up time (TBUT) from baseline to Day 0 (surgical day) and Day 7 to Day 28 (1-month postoperative CXL)
Adverse Events | 56 days (4 weeks preop and 4 weeks postop)
  Incidence and severity of adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Vance Thompson Vision-MT, Bozeman, Montana, United States

REFERENCES:
- [Derived] Ferguson TJ, Durgan D, Whitt T, Swan RJ. Varenicline Nasal Spray for the Treatment of Dry Eye Disease Following Corneal Collagen Crosslinking. Ophthalmol Ther. 2025 May;14(5):959-968. doi: 10.1007/s40123-025-01118-x. Epub 2025 Mar 15. PMID 40088395